CLINICAL TRIAL: NCT03638843
Title: Endoscopic Gastric Mucosal Devitalization (GMD) as a Primary Obesity Therapy - Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00089675-2
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Obesity, Morbid; Obesity; Endocrine; Bariatric Surgery Candidate
Keywords: bariatric endoscopy; obesity; metabolic syndrome; gastric mucosal devitalization; Endoscopic bariatric therapies
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric mucosal devitalization arm (Experimental): Patients will be enrolled in the study after being scheduled to undergo vertical sleeve gastrectomy as part of routine clinical care, and the gastric mucosal devitalization procedure will be performed in-vivo utilizing Argon plasma coagulation three days before the operation.
  Interventions: Procedure: Gastric mucosal devitalization

INTERVENTIONS:
Procedure: Gastric mucosal devitalization — Gastric mucosal devitalization is an endoscopic procedure which uses argon plasma coagulation to result in selective damage to the gastric mucosa and submucosa.

SUMMARY:
Rapid metabolic improvements seen with sleeve gastrectomy are likely a result of changes in gastric origin. The gastric mucosa is an endocrine organ that regulates satiation pathways and is a complex regulator of food intake as well as lipid and glucose metabolism. This study aims to assess the efficacy and safety of endoscopic selective gastric mucosal devitalization (GMD) for the management of obesity and its related comorbidities.

DETAILED DESCRIPTION:
Endoscopic approaches to obesity may help fulfill the unmet need of over half the US adult population that would benefit from therapy for obesity but are not receiving it. Endoscopic approaches to obesity have the potential to be more efficacious than antiobesity medications and have a lower risk-cost profile compared with bariatric surgery.

Endoscopic approaches to obesity need to be increasingly modeled on the proposed mechanisms contributing to the benefits of bariatric surgery.

The investigators seek to decipher if the gastric mucosa is an independent regulator of food intake, body weight, lipid and glucose metabolism and serum gut hormones. The investigators also wish to ascertain if selective devitalization of the gastric mucosa, without alteration in gastric volume, will improve obesity related comorbidities.

This study will be divided into 3 parts. The purpose of completing the 3 phases is to develop a minimally invasive weight loss technique that is effective, safe and ready for more rigorous assessment via a future randomized control trial.

Objectives:

Overall:

To assess the efficacy and safety of gastric mucosal devitalization for the management of obesity and its related comorbidities.

Part 2:

Aims to confirm that the optimal color of the tissue identified by part 1 corresponds to selective mucosal devitalization in the in vivo setting by histopathologic examination. For this, patients will be enrolled in the study after being scheduled to undergo vertical sleeve gastrectomy (VSG). GMD will be performed three days prior to the VSG, and the excised tissue including devitalized gastric mucosa will be evaluated. The degree and correlation of devitalization with mucosal discoloration will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo vertical sleeve gastrectomy

Exclusion Criteria:

* Age under 28 or older than 60
* Insulin dependent Diabetes Mellitus
* Suspected or biopsy confirmed liver cirrhosis
* Significant ethanol consumption >21 drinks/week in men and >14 drinks/week in women
* Presence of other chronic liver disease including hepatitis B-C, autoimmune hepatitis, alpha 1 antitrypsin deficiency, Wilson's disease, and hemochromatosis
* Pregnant or breast-feeding
* Patients who already have an intragastric balloon or other gastric implant
* Patients with gastroesophageal reflux disease
* Patients with previous gastric surgeries, altered gastrointestinal anatomy such as Billroth I, Billroth II, roux-en-y gastrectomy, roux-en-y hepaticojejunostomy, or any restrictive or bypass bariatric surgery
* Patients with previous gastric embolization for obesity
* Presence of inflammatory disorder of the gastrointestinal tract
* Patients with active peptic ulcer disease
* Patients with gastroesophageal varices
* Presence of a large hiatal hernia (grade IV on Hills classification: large hiatal hernia and essentially no fold approximating the endoscope in the retroflexed view and where the lumen of the esophagus is gaping open allowing the squamous epithelium to be seen)
* Structural abnormality in the esophagus or pharynx
* Have major esophageal motility disorders as per the Chicago classification including achalasia, diffuse esophageal spasm, jackhammer esophagus, and Esophagogastric junction outflow obstruction
* Mucosal or submucosal gastric mass that is clinically suspected to be of malignant nature
* Severe clotting or bleeding disorder
* Other medical condition that does not allow for endoscopic procedure
* Severe psychiatric illness
* Unable to participate in routine medical follow-up
* On antiplatelet agents including clopidogrel, ticlopidine, prasugrel, and cangrelor. acetylsalicylic acid use will be allowed
* On anticoagulants including heparin, warfarin, dabigatran, rivaroxaban, apixaban, and edoxaban

Ages: 28 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Pathological changes | 6 months
  Histopathological assessment to determine whether selective devitalization of mucosa and submucosa corresponds with decolorization during the in-vivo procedure.

SECONDARY OUTCOMES:
Technical feasibility | 6 months
  Feasibility of retroflexion technique during the in-vivo devitalization procedure assessed by the endoscopist.
Procedural tolerability | 6 months
  Tolerability of gastric mucosal devitalization after the post-procedural follow up assessed by the endoscopist

CONTACTS AND LOCATIONS:
Overall Officials: Dilhana Badurdeen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States